CLINICAL TRIAL: NCT06652126
Title: Impact of Immunosuppression on Intensive Care Unit-acquired Multidrug-resistant Bacteria: a Prospective Multicenter Study in Europe
Brief Title: Immunosuppression and Intensive Care Unit-acquired Multidrug-resistant Bacteria
Acronym: TANGERINE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_0226; 2023-A02489-36 (Other: ID-RCB Number)
Record Dates: First submitted 2024-09-23; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Critically-ill Patients
Keywords: Immunocompromised patients; antimicrobial resistance; intensive care unit; cross-infections
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunocompromised patients: * Age ≥ 18 ;
  * Admitted to intensive care and whose length of stay exceeds 48 hours ;
  * Immunocompromised according to one of the following criteria:
    1. Solid cancer under treatment or in remission for less than 5 years (including cancers diagnosed during hospitalization in intensive care) ;
    2. Hematologic malignancy under treatment or in remission for less than 5 years (including hematologic malignancies diagnosed during hospitalization in intensive care);
    3. Neutropenia < 0.7 G/L for ≥ 7 days;
    4. Solid organ transplants;
    5. Patients with systemic or transplant pathologies requiring treatment with corticosteroids (prednisone equivalent > 10 mg/day) or other high-dose immunosuppressants for > 28 days;
    6. Human Immunodeficiency Virus (HIV) infection with CD4+ <200 μL;
    7. Genetic immune deficiency.
  * Undergoing invasive mechanical ventilation and/or vasopressive amines.
  Interventions: Other: Microbiological examinations.
- Immunocompetent patients: * Age ≥ 18 ;
  * Admitted to intensive care and whose length of stay exceeds 48 hours ;
  * Immunocompetent ;
  * Undergoing invasive mechanical ventilation and/or vasopressive amines.
  Interventions: Other: Microbiological examinations.

INTERVENTIONS:
Other: Microbiological examinations. — * BMR testing by rectal swab (combined with nasal swab in some centers) on admission to the ICU and weekly as part of routine care.
  * Microbiological samples (blood cultures, respiratory and urinary samples, etc.) as part of routine care at the request of the clinicians in charge of the patient.

SUMMARY:
Antimicrobial resistance AMR is an emerging global threat to human health, and intensive care units (ICUs) are a 'hot spot' for the emergence and diffusion of multidrug-resistant (MDR) bacteria. ICU-acquired colonization and infection with MDR bacteria (ICU-MDR-col and ICU-MDR-inf, respectively) have been associated with higher ICU length-of-stay, duration of invasive mechanical ventilation and mortality. Immunocompromised patients account for an increasing proportion of ICU patients, and they are particularly prone to ICU-acquired infections, a significant proportion of which are caused by MDR pathogens. Recently, in a prospective multicenter study in France (CIMDREA, 8 ICUs, 750 patients), we found that immunocompromised patients had a lower cumulative incidence of ICU-MRD-col, but not ICU-MDR-inf (after adjustment for confounders). These results suggest that isolation measures and contact precautions could have a protective impact on cross-transmission of MDR bacteria in immunocompromised patients, even though our study fails to provide conclusive arguments for this. If confirmed, these findings could have an impact on antibiotic stewardship in immunocompromised critically-ill patients, a key element to control the spread of AMR in ICUs and beyond. Thus, we are planning to carry out the TANGERINE study, an observational prospective multicenter study in Europe, to confirm the findings of CIMDREA and provide a better understanding of the effect of isolation measures and contact precautions on the epidemiology of AMR in ICUs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 and over.
2. Admitted to intensive care and whose length of stay is greater than 48 hours (inclusion is at the 48th hour after admission).
3. Immunocompetent OR immunocompromised patients according to one of the following criteria:

   1. Solid cancer under treatment or in remission for less than 5 years (including cancers diagnosed during hospitalization in intensive care);
   2. Hematological malignancies under treatment or in remission for less than 5 years (including hematological malignancies diagnosed during hospitalization in intensive care);
   3. Neutropenia < 0.7 G/L for ≥ 7 days;
   4. Solid organ transplants;
   5. Patients with systemic or transplant pathologies requiring treatment with corticosteroids (prednisone equivalent > 10 mg/day) or other high-dose immunosuppressants for > 28 days;
   6. Human Immunodeficiency Virus (HIV) infection with CD4+ <200 μL;
   7. Genetic immune deficiency.
4. Patients undergoing invasive mechanical ventilation and/or vasopressive amines.
5. Persons who have given their non-opposition. For patients unable to give their non-opposition, this will be obtained from the trusted support person. The patient will be informed as soon as possible and asked to agree to participate in any further research.
6. Patients affiliated to a social security system.

Exclusion Criteria:

1. Minor patients (< 18 years),
2. Length of stay in intensive care less than 48 hours,
3. Moribund patients.
4. Absence of BMR screening (rectal swab routinely, combined with nasal swab in some centers) within 48 hours of admission.
5. Refusal to participate in the study.
6. Vulnerable and/or susceptible patients according to one of the following criteria:

   1. Patients under legal protection (guardianship, curatorship, etc.);
   2. Patients in prison;
   3. Pregnant or breast-feeding women.
7. Patients without social security coverage.
8. Simultaneous participation in another interventional study that could interfere with the evaluation of primary and secondary endpoints (particularly in the case of participation in an interventional study that could modulate the risk of CAR or BMR-ARI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care units (ICU).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare the 28-day cumulative incidence of a composite outcome including ICU-MDR-col and/or ICU-MDR-inf between immunocompromised and non-immunocompromised patients. | End of ICU-stay or day 28 after ICU admission (whichever comes first)

SECONDARY OUTCOMES:
To compare the 28-day cumulative incidence of ICU-MDR-col between immunocompromised and non-immunocompromised patients. | End of ICU-stay or day 28 after ICU admission (whichever comes first)
To compare the 28-day cumulative incidence of ICU-MDR-inf between immunocompromised and non-immunocompromised patients. | End of ICU-stay or day 28 after ICU admission (whichever comes first)
To compare the incidence rate of a composite outcome including ICU-MDR-col and/or ICU-MDR-inf between immunocompromised and non-immunocompromised patients. | End of ICU-stay or day 28 after ICU admission (whichever comes first)
To compare the incidence rate of ICU-MDR-col between immunocompromised and non-immunocompromised patients. | End of ICU-stay or day 28 after ICU admission (whichever comes first)
To compare the incidence rate of ICU-MDR-inf between immunocompromised and non-immunocompromised patients. | End of ICU-stay or day 28 after ICU admission (whichever comes first)
To evaluate the effect of contact precautions and isolation measures on the 28-day cumulative incidence of ICU-MDR-col and ICU-MDR-inf in immunocompromised patients. | End of ICU-stay or day 28 after ICU admission (whichever comes first)
To describe the microbiology of ICU-MDR-col and ICU-MDR-inf in immunocompromised and non-immunocompromised patients | End of ICU-stay or day 28 after ICU admission (whichever comes first)
To assess the effect of the type of immunosuppression on the 28-day cumulative incidence of ICU-MDR-col and ICU-MDR-inf among immunocompromised patients. | End of ICU-stay or day 28 after ICU admission (whichever comes first)
To evaluate the association of occurrence of ICU-MDR-col and ICU-MDR-inf and prognostic outcomes (ICU length-of-stay, duration of IMV and 28-day mortality) in the overall cohort and according to immune status (i.e., in immunocompromised and non-immunocom | End of ICU-stay or day 28 after ICU admission (whichever comes first)

IPD SHARING:
Plan to Share IPD: No